CLINICAL TRIAL: NCT02746029
Title: Cardiac Murmurs in Children: Predictive Value of Cardiac Markers
Acronym: CAMUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Wyller, Professor, University Hospital, Akershus
Other Study IDs: CAMUS
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with cardiac murmur
  Interventions: Other: Clinical examination

INTERVENTIONS:
Other: Clinical examination

SUMMARY:
Heart murmurs are commonly discovered in young children during clinical encounters in general practice. Heart murmurs might signal a structural cardiac disease that need to be treated, such as atrial septal defect. Thus, children with heart murmurs are routinely referred to comprehensive cardiac examination at a paediatric hospital department featuring echocardiography ('gold standard'). However, the great majority of such murmurs are innocent or physiological; ie., they do not represent a cardiac disorder. The prevalence of such innocent murmurs during routine random auscultation is estimated at 30 %.

It would be advantageous if patients with a heart disease to a greater extent could be identified at the general practitioners' office:

* Healthy children would not be exposed to comprehensive cardiac examination
* The burden on the family would subside.
* Scarce medical resources in highly specialized departments would be better allocated, to the benefit of patients with real heart disease.

The primary aim of this study is to establish the predictive value of cardiac markers in children with heart murmurs. Secondary aims are a) To do a pilot study of pediatric cardiac ultrasound examination in general practice; b) To establish age-adjusted reference range for cardiac markers in children, and c) To explore aspects of cardiovascular physiology in children.

The investigators will include a total of 500 children aged 4 weeks to 10 years who is consecutively referred to the Dept. of Paediatrics, Akershus University Hospital, for assessment of heart murmurs. All participants will be subjected to clinical examination, symptom assessment, pulse oximetry, blood sampling (for troponin T, proBNP and other biomarkers), ECG recording, and echocardiography. A randomized subgroup of children will also undergo echocardiography performed by a general practitioner who has not received formal training in pediatric cardiology. The value of possible predictors will be assessed through the construction of Receiver Operating Characteristics (ROC) curves, and calculation of negative predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneously discovered heart murmur at general practitioner's office

Exclusion Criteria:

* Known cardiac disease
* Other chronic or acute disorder
* Medications

Ages: 4 Weeks to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children consecutively referred to Akerhus University Hospital for spontaneously discovered cardiac murmur in general practice.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with any congenital heart disease as assessed by echocardiography | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Wyller, Principal Investigator — University Hospital, Akershus
Locations (1):
- Dept. of Pediatrics, Akershus University Hospital, Lørenskog, Akershus, Norway

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT02746029/SAP_000.pdf